CLINICAL TRIAL: NCT04379050
Title: An Open-label Extension of Study M15-741 to Evaluate the Safety and Tolerability of 24-hour Daily Exposure of Continuous Subcutaneous Infusion of ABBV-951 in Subjects With Parkinson's Disease
Brief Title: Extension Study To Evaluate Safety And Tolerability Of 24-Hour Daily Exposure Of Continuous Subcutaneous Infusion of ABBV-951 In Adult Participants With Parkinson's Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-737; 2019-004235-23 (EudraCT Number)
Record Dates: First submitted 2020-05-01; First posted 2020-05-07 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's Disease (PD); ABBV-951; Levodopa/Carbidopa (LD/CD); Levodopa Phosphate/Carbidopa Phosphate (LDP/CDP)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ABBV-951 (Experimental): Participants will receive ABBV-951 solution by continuous subcutaneous infusion (CSCI), at the discretion of the investigator, for up to 96 weeks.
  Interventions: Drug: ABBV-951

INTERVENTIONS:
Drug: ABBV-951 — Solution for continuous subcutaneous infusion (CSCI).
  Other Names: Foscarbidopa; Foslevodopa

SUMMARY:
Parkinson's disease (PD) is a neurological condition, which affects the brain. PD gets worse over time, but how quickly it progresses varies a lot from person to person. Some symptoms of PD are tremors, stiffness, and slowness of movement. The purpose of this study is to continue testing whether ABBV-951 is safe, effective, and tolerable in participants with Parkinson's disease after completion of the parent study M15-741.

ABBV-951 is an investigational (unapproved) drug containing levodopa phosphate/carbidopa phosphate (LDP/CDP) given as infusion under the skin for the treatment of Parkinson's Disease. Participants who have successfully completed M15-741 study will immediately enter this study's treatment period to continue receiving ABBV-951. Adult participants with advanced PD will be enrolled. Approximately 130 adult participants will be enrolled in the study at approximately 65 sites worldwide.

Participants will receive continuous subcutaneous infusion (CSCI) of ABBV-951 for 24 hours daily during the Primary Treatment Period and during the optional Extended Treatment Period.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular clinic visits and have remote assessments completed via phone calls during the course of the study. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have Parkinson's Disease and who have successfully completed the parent study M15-741.
* Participants willing and able to comply with procedures required in the protocol.

Exclusion Criteria:

- Participants, if judged by the investigator to be unsuitable candidates to continue to receive ABBV-951 for any reason.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AE) | Up To Week 96
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of the study drug or device as either reasonable possibility or no reasonable possibility. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Adverse Events of Special Interest (AESI) - polyneuropathy, weight loss, hallucinations/psychosis, and somnolence will be monitored throughout the study.
Percentage Of Participants With Numeric Grade Equal To Or Higher Than 5 On The Infusion Site Evaluation Scale | Up To Week 96
  The Infusion Site Evaluation Scale will be used to assess infusion sites. Infusion Site Evaluation Scale is an eight-point numeric scale used to assess irritation at the infusion site area (0 being "no evidence of irritation" and 7 being "strong reaction spreading beyond the test site").
Percentage Of Participants With Letter Grade Equal To Or Higher Than D On The Infusion Site Evaluation Scale | Up To Week 96
  The Infusion Site Evaluation Scale will be used to assess infusion sites. Infusion Site Evaluation Scale is an A to G letter grade scale, used to assess irritation at the infusion site area (A being "no finding" to G being "Small petechial erosions and/or scabs").
Change in Clinical Laboratory Test Data | Up To Week 96
  Number of participants with clinically significant change from baseline in laboratory parameters (hematology, biochemistry, coagulation, and urinalysis) will be reported throughout the study.
Change in Vital Signs Measurements | Up To Week 96
  Number of participants with clinically significant change from baseline in vital signs will be reported throughout the study.
Change From Baseline in Electrocardiograms (ECGs) | Up To Week 96
  Change from baseline in 12-lead ECGs on heart rate, RR interval, PR interval, QRS duration, and QT interval will be monitored throughout the study.

SECONDARY OUTCOMES:
Average Normalized Daily "Off" Time | Up To Week 96
  Average normalized daily "Off" Time (Hours) is assessed based on Parkinson's Disease (PD) Diary.
Average Normalized Daily "On" Time | Up To Week 96
  Average normalized daily "On" time is assessed based on Parkinson's Disease (PD) Diary.
Parkinson's Disease (PD) Symptoms Measurement | Up To Week 96
  PD symptoms will be assessed by the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I-IV.
  The MDS-UPDRS is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD) with scores ranging from 0 to 236 with 236 representing the worst disability, and 0 representing no disability.
Change From Baseline in Quality Of Life Measurement as Assessed by PD Questionnaire-39 (PDQ-39) | Up To Week 96
  Quality of life is assessed by the PD Questionnaire-39 items (PDQ-39). PDQ-39 is a disease-specific instrument designed to measure aspects of health that are relevant to participants with PD, and which may not be included in general health status questionnaires.
  Each item is scored on a 5-point scale.
Change From Baseline in Health-related Quality Of Life Measurement as Assessed by EuroQol 5-dimensions questionnaire (EQ-5D-5L) | Up To Week 96
  Health-related quality of life is assessed by the EuroQol 5-dimensions questionnaire (EQ-5D-5L).
  EQ-5D-5L is a standardized instrument that consists of 2 parts: the EQ-5D descriptive system and the EQ visual analogue-scale (EQVAS).
Cognitive Impairment Measurement | Up To Week 96
  Cognitive impairment is assessed by the Mini-Mental State Examination (MMSE). MMSE is used to assess orientation, attention, immediate and short term recall, language, and ability to follow simple verbal and written commands. The test consists of five sections (orientation, registration, attention-calculation, recall, and language) and results in a total possible score of 0 to 30, with higher scores indicating better function.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (51):
- United States (15):
  - University of Alabama at Birmingham - Main /ID# 215597, Birmingham, Alabama
  - Banner Sun Health Research Institute /ID# 215579, Sun City, Arizona
  - University of Colorado Hospital /ID# 215625, Aurora, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton /ID# 215412, Boca Raton, Florida
  - Indiana Clinical Research Cent /ID# 216490, Indianapolis, Indiana
  - Univ Kansas Med Ctr /ID# 215624, Kansas City, Kansas
  - Washington University-School of Medicine /ID# 215472, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center /ID# 216834, Lebanon, New Hampshire
  - M3 Wake Research Inc. /ID# 215596, Raleigh, North Carolina
  - Legacy Medical Group - Neurology /ID# 215536, Portland, Oregon
  - Baylor College of Medicine /ID# 215401, Houston, Texas
  - Central Texas Neurology Consul /ID# 217013, Round Rock, Texas
  - Univ Texas HSC San Antonio /ID# 215400, San Antonio, Texas
  - Booth Gardner Parkinson's Care Center /ID# 215535, Kirkland, Washington
  - Inland Northwest Research /ID# 215533, Spokane, Washington
- Australia (5):
  - Concord Repatriation General Hospital /ID# 215943, Concord, New South Wales
  - Westmead Hospital /ID# 215941, Westmead, New South Wales
  - Duplicate_Royal Adelaide Hospital /ID# 215940, Adelaide, South Australia
  - The Alfred Hospital /ID# 215942, Melbourne, Victoria
  - Perron Institute /ID# 215944, Nedlands, Western Australia
- Belgium (3):
  - Universitair Ziekenhuis Leuven /ID# 215684, Leuven, Vlaams-Brabant
  - Duplicate_Algemeen Ziekenhuis Sint-Jan Brugge /ID# 215686, Bruges, West-Vlaanderen
  - Duplicate_Groupe Sante CHC - Clinique du MontLegia /ID# 215685, Liège
- Canada (2):
  - University of Calgary /ID# 215369, Calgary, Alberta
  - Clinique Neuro Levis /ID# 215371, Lévis, Quebec
- Denmark (3):
  - Bispebjerg and Frederiksberg Hospital /ID# 215391, Copenhagen NV, Capital Region
  - Aarhus Universitetshospital - Skejby /ID# 215392, Aarhus, Central Jutland
  - Odense University Hospital /ID# 215390, Odense, Region Syddanmark
- Germany (3):
  - Universitaetsklinikum Ulm /ID# 215405, Ulm, Baden-Wurttemberg
  - curiositas ad sanum /ID# 215404, Haag i.OB, Bavaria
  - Kliniken Beelitz GmbH /ID# 215403, Beelitz-Heilstätten
- Italy (2):
  - IRCCS Centro Neurolesi Bonino Pulejo /ID# 215422, Messina
  - Azienda Ospedale-Universita Padova /ID# 215421, Padua
- Japan (3):
  - National Hospital Organization Asahikawa Medical Center /ID# 218762, Asahikawa-shi, Hokkaido
  - Duplicate_Osaka University Hospital /ID# 217415, Suita-shi, Osaka
  - National Center of Neurology and Psychiatry /ID# 218763, Kodaira-shi, Tokyo
- St. Antonius Ziekenhuis /ID# 215396, Nieuwegein, Utrecht, Netherlands
- Russia (2):
  - Academician I.P. Pavlov First St. Petersburg State Medical University /ID# 218869, Saint Petersburg, Sankt-Peterburg
  - City Clinical Hospital #40 /ID# 218870, Sestroretsk, Sankt-Peterburg
- Spain (6):
  - Complejo Hospitalario Universitario A Coruña /ID# 215426, A Coruña, A Coruna
  - Hospital General Universitario de Elche /ID# 215425, Elche, Alicante
  - Hospital Universitari de Bellvitge /ID# 215427, L'Hospitalet de Llobregat, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 215429, Barcelona
  - Hospital Universitario Virgen de las Nieves /ID# 215431, Granada
  - Hospital Universitario Virgen del Rocio /ID# 215428, Seville
- Sweden (3):
  - Skane University Hospital Lund /ID# 215385, Lund, Skåne County
  - Karolinska Universitetssjukhuset - Huddinge /ID# 215386, Huddinge, Stockholm County
  - Sahlgrenska Universitetssjukhuset /ID# 215387, Gothenburg, Västra Götaland County
- United Kingdom (3):
  - Derriford Hospital and the Royal Eye Infirmary /ID# 217390, Plymouth, Devon
  - NHS Tayside /ID# 217389, Dundee, Scotland
  - King's College Hospital NHS Foundation Trust /ID# 217388, London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/